CLINICAL TRIAL: NCT06798064
Title: Expanded Access Using Allogeneic Bone-marrow Derived Human Mesenchymal Stem Cells (Allo-hMSC) for a Individual Parkinson's Disease Subject
Status: No longer available | Type: Expanded Access
Sponsor: Mya Schiess (Other)
Responsible Party: Sponsor-Investigator, Mya Schiess, Professor, The University of Texas Health Science Center, Houston
Organization: The University of Texas Health Science Center, Houston (Other)
Other Study IDs: HSC-MS-24-1279
Record Dates: First submitted 2025-01-16; First posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Biological: Allogeneic bone marrow-derived mesenchymal stem cells

SUMMARY:
This is a expanded access use of allogeneic bone marrow-derived mesenchymal stem cells for a single subject with moderate Parkinson's disease that has progressed.

Ages: 50 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Mya Schiess, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States